CLINICAL TRIAL: NCT00624572
Title: Efficacy of 1% Chlorexidine Gel as Intracanal Medicament in Primary Molar Teeth - a Clinical and Microbiological Study
Brief Title: Efficacy of Chlorexidine as Intracanal Medicament in Primary Teeth
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Federal do Ceara (Other)
Responsible Party: Ramille Araújo Lima, Federal University of Ceará
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CHX0784
Record Dates: First submitted 2008-02-15; First posted 2008-02-27 (Estimated); Last update posted 2008-02-27 (Estimated); Status verified 2008-02

CONDITIONS: Dental Pulp Necrosis
Keywords: primary teeth; chlorexidine; root canal therapy; Pulpectomy
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Drug: chlorexidine — Chlorexidine gel 1% during 7 days inside root canals

SUMMARY:
The purpose of this study is to evaluate the action of the chlorexidine as intracanal medicament in the reduction of the levels of bacteria inside root canals of primary molar teeth with pulpal necrosis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children of both gender;
* Without history of reactions or alergical diseases;
* With situated age between 04 and 08 years of age
* With normal standard of growth and development
* Patients with necessity of radical endodontic treatment (pulpectomy) in, at least, two primary molar teeth in different hemi-arches.

Exclusion Criteria:

* Patients with history of alergical diseases
* Patients with allergy to any type of medicine and/or foods
* Patients with comprometimento of its general state of health
* Healthy patients with risk to develop bacterial endocardite or patients that their general state of health can be aggravated had the transitory bacteremies, as for example children with congenital cardiac illnesses
* Patients who are making use of sistemis antibiotics, or that they have made use of sistemic antibiotic in the period of 3 (three) months before the beginning of the endodontic treatment
* With periapical x-ray evidencing less than 2/3 of remaining root of the primary tooth to be treated
* Patients whose tooth with endodontic necessity to meet in advanced state of root pathological reabsortion
* Patients whose legal responsible or parents to refuse to sign the term of free and clarified assent

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-11 (Estimated); Study Completion 2009-02 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Ramille Araújo Lima, Fortaleza, Ceará, Brazil